CLINICAL TRIAL: NCT06685276
Title: A Prospective Single-arm Phase Ib/II Study on the Safety and Efficacy of Fruquintinib Plus Chidamide and Sintilimab in the Third and Later Line Treatment of MSS/pMMR Metastatic Colorectal Cancer
Brief Title: Safety and Efficacy of Fruquintinib Plus Chidamide and Sintilimab in the Third and Later Line Treatment of MSS/pMMR Metastatic Colorectal Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Dai, Guanghai (Other)
Responsible Party: Sponsor-Investigator, Dai, Guanghai, Chief Physician, Chinese PLA General Hospital
Organization: Chinese PLA General Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-415
Record Dates: First submitted 2024-11-11; First posted 2024-11-12 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Colorectal Cancer Metastatic
MeSH Terms: interventions — HMPL-013; sintilimab; N-(2-amino-5-fluorobenzyl)-4-(N-(pyridine-3-acrylyl)aminomethyl)benzamide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Study arm (Experimental): Fruquintinib Sintilimab Chidamide
  Treatments are administered until disease progression or toxicity intolerable.
  Interventions: Drug: Fruquintinib; Drug: Sintilimab; Drug: Chidamide

INTERVENTIONS:
Drug: Fruquintinib — Fruquintinib: 5mg qd, po, 2 weeks on/1 week off, q3w, or 3mg qd, po, q3w.
  Other Names: hmpl-013
Drug: Sintilimab — Sintilimab: 200mg, iv, d1, q3w.
Drug: Chidamide — Chidamide: 30mg/m2, po, biw.

SUMMARY:
The prognosis of most patients with unresectable locally advanced or metastatic colorectal cancer (CRC) remains poor despite the advancements in chemotherapy and target therapy.

CAPability-01 trial investigated the potential efficacy of combining the programmed cell death protein-1 (PD-1) monoclonal antibody sintilimab with the histone deacetylase inhibitor (HDACi) chidamide with or without the anti-vascular endothelial growth factor (VEGF) monoclonal antibody bevacizumab in patients with unresectable chemotherapy-refractory locally advanced or metastatic microsatellite stable/proficient mismatch repair (MSS/pMMR) colorectal cancer.

Based on the previous findings of CAPability-01, we will further evaluate the efficacy and safety of sintilimab and chidamide in combination with fruquintinib in the same setting.

ELIGIBILITY:
Inclusion Criteria:

1. Fully understand this study and voluntarily sign the informed consent form;
2. Age between 18-75 years inclusive;
3. Patients with histologically confirmed unresectable locally advanced, recurrent, or metastatic colorectal adenocarcinoma;
4. Failure of standard second-line systemic treatment with measurable lesions;
5. Tumor tissue tested for microsatellite stability (MSS) or low microsatellite instability (MSI-L) by PCR, or confirmed pMMR by immunohistochemistry for DNA mismatch repair (MMR) protein (including MLH1, MSH2, MSH6, and PMS2 protein expression);
6. ECOG performance status of 0-2, with no deterioration within 7 days;
7. BMI≥18;
8. Expected survival ≥3 months;
9. Major organ functions meet the following requirements (no use of any blood components and growth factors within 14 days before enrollment):

   * Absolute neutrophil count ≥1.5×109/L, white blood cells ≥4.0×109/L;
   * Platelets ≥100×109/L;
   * Hemoglobin ≥90g/L;
   * Total bilirubin TBIL ≤1.5 times ULN;
   * ALT and AST ≤5 times ULN;
   * Urea/BUN and creatinine (Cr) ≤1.5×ULN (and creatinine clearance (CCr) ≥ 50mL/min);
   * Left ventricular ejection fraction (LVEF) ≥50%;
   * Corrected QT interval by Fridericia's formula (QTcF) <470 milliseconds.
   * INR ≤1.5×ULN, APTT ≤1.5×ULN.
10. Women of childbearing age must use effective contraception;
11. Good compliance and cooperation with follow-up.

Exclusion Criteria:

1. Unable to comply with the study protocol or procedures;
2. Pregnant or breastfeeding women;
3. Concurrent with any of the following conditions: uncontrolled hypertension, coronary artery disease, arrhythmias, and heart failure;
4. Previous treatment with small molecule tyrosine kinase inhibitors for metastatic disease;
5. Previous treatment with romidepsin;
6. Previous treatment with immune checkpoint inhibitors for metastatic disease;
7. Uncontrollable severe concurrent infections;
8. Acute myocardial infarction, acute coronary syndrome, or CABG within 3 months before the first treatment;
9. Subjects allergic to the study medication or any of its excipients;
10. Known human immunodeficiency virus (HIV) infection. Known clinically significant liver disease history, including viral hepatitis [known carriers of hepatitis B virus (HBV) must exclude active HBV infection, i.e., HBV DNA positive (>1×10^4 copies/mL or >2000 IU/mL); known hepatitis C virus (HCV) infection and HCV RNA positive (>1×10^3 copies/mL)];

12. Patients whom the investigator deems inappropriate for inclusion in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2024-08-16 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Progress-free Survival(PFS) | 24 months
  The time from enrollment until tumor progression or death from any cause, whichever occurred first

SECONDARY OUTCOMES:
Objective response rate (ORR) | 24 months
  The proportion of patients with a PR or CR
Overall Survival (OS) | 24 months
  The time calculated from enrollment until death from any cause, with living patients censored at the last known survival date
Disease control rate (DCR) | 24 months
  The proportion of patients with a PR, CR, or SD
Duration of response (DoR) | 24 months
  For patients who achieved a complete response (CR) or partial response (PR), the time from the first tumor assessment demonstrating response until disease progression or death, whichever occurred first

CONTACTS AND LOCATIONS:
Locations (1):
- China PLAGH, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided